CLINICAL TRIAL: NCT03228732
Title: The Effects of the Selective Serotonin Reuptake Inhibitor, Fluoxetine and/or DHEA, on Neuroendocrine, Autonomic Nervous System and Metabolic Counterregulatory Responses During Repeated Hypoglycemia in T1DM Individuals
Brief Title: The Effects of Fluoxetine and/or DHEA
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Stephen N. Davis, MBBS, Chairman of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HP-00075896
Record Dates: First submitted 2017-07-20; First posted 2017-07-25 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Fluoxetine; Dehydroepiandrosterone

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 2 groups. Group 1 will consist of a random order of Protocol 1 and Protocol 5. Group 2 will consist of a randomized order of Protocols 2, 3, 4
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo 1 (Placebo Comparator): Visit 1:
  Study Day 1: Hyperinsulinemia/ euglycemia clamp in the AM and PM. Study Day 2: Hyperinsulinemia/ hypoglycemia clamp in the AM only. 8-weeks of treatment with placebo
  Visit 2:
  same as visit 1
  Interventions: Drug: Placebo Oral Tablet
- Placebo 2 (Placebo Comparator): Visit 1:
  Study Day 1: Hyperinsulinemia/ hypoglycemia clamp in the AM and PM. Study Day 2: Hyperinsulinemia/ hypoglycemia clamp in the AM only. 8-weeks of treatment with placebo
  Visit 2:
  same as visit 1
  Interventions: Drug: Placebo Oral Tablet
- Fluoxetine (Active Comparator): Visit 1:
  Study Day 1: Hyperinsulinemia/ hypoglycemia clamp in the AM and PM. Study Day 2: Hyperinsulinemia/ hypoglycemia clamp in the AM only. 8-weeks of treatment with fluoxetine
  Visit 2:
  same as visit 1
  Interventions: Drug: Fluoxetine
- DHEA (Active Comparator): Visit 1:
  Study Day 1: Hyperinsulinemia/ hypoglycemia clamp in the AM and PM. Study Day 2: Hyperinsulinemia/ hypoglycemia clamp in the AM only. 8-weeks of treatment with DHEA
  Visit 2:
  same as visit 1
  Interventions: Drug: DHEA
- Fluoxetine and DHEA (Active Comparator): Visit 1:
  Study Day 1: Hyperinsulinemia/ hypoglycemia clamp in the AM and PM. Study Day 2: Hyperinsulinemia/ hypoglycemia clamp in the AM only. 8-weeks of treatment with fluoxetine and DHEA
  Visit 2:
  same as visit 1
  Interventions: Drug: Fluoxetine and DHEA

INTERVENTIONS:
Drug: Placebo Oral Tablet — There will be two 2-day inpatient visits with 8-weeks of treatment with placebo between those visits.
  Arms: Placebo 1
Drug: Placebo Oral Tablet — There will be two 2-day inpatient visits with 8-weeks of treatment with placebo between those visits.
  Arms: Placebo 2
Drug: Fluoxetine — There will be two 2-day inpatient visits with 8-weeks of treatment with fluoxetine between those visits.
  Arms: Fluoxetine
Drug: DHEA — There will be two 2-day inpatient visits with 8-weeks of treatment with DHEA between those visits.
  Other Names: dehydroepiandrosterone
  Arms: DHEA
Drug: Fluoxetine and DHEA — There will be two 2-day inpatient visits with 8-weeks of treatment with fluoxetine and DHEA between those visits.
  Other Names: Prozac, dehydroepiandrosterone
  Arms: Fluoxetine and DHEA

SUMMARY:
(1) To determine how the Selective Serotonin Reuptake Inhibitor (SSRI), fluoxetine (Prozac), an antidepressant often used to treat depression, stimulates the participant's body's ability to defend against low blood sugar (hypoglycemia). (2) To learn how a hormone, dehydroepiandrosterone (DHEA), stimulates the participant's body's ability to defend itself from low blood sugar (hypoglycemia). DHEA is a hormone produced naturally in the human body. However, it can be manufactured and is sold as an over-the-counter dietary supplement. The dose the investigators are giving in this study is higher than the usual recommended dosage taken as a supplement for certain medical conditions. (3) To study combined effects of fluoxetine and DHEA during low blood glucose. In the present study, the investigators will measure the participant's body's responses to hypoglycemia when given fluoxetine or DHEA or fluoxetine and DHEA or a placebo (a pill with no fluoxetine or DHEA). Approximately 64 individuals with type 1 diabetes will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* 64 (32 males, 32 females) T1DM patients aged 18-50 yr.
* HbA1c < 11.0%
* No clinically diagnosed diabetic tissue complications (i.e. history of retinopathy, neuropathy, stasis ulcers, etc)
* Body mass index < 40kg · m-2

Exclusion Criteria:

* Pregnancy
* Subjects unable to give voluntary informed consent
* Subjects on anticoagulant drugs, anemic or with known bleeding diatheses
* Subjects taking any of the following medications will be excluded: Non-selective Beta Blockers, Sedative-Hypnotics, Anticonvulsants, Antiparkinsonian drugs, Antipsychotics, Antidepressants, Mood stabilizers, CNS Stimulants, Opioids, Hallucinogens
* Subjects with a recent medical illness or past history of severe depression, mania or psychotic disease
* Subjects that score greater than 50 on the depression scale
* Subjects unwillingness or inability to comply with approved contraception measures
* Abnormal results following screening tests and physical examination that are clinically significant
* Subjects with a history of severe uncontrolled hypertension (i.e., blood pressure greater than 160/100), heart disease, cerebrovascular incidents
* Clinically significant cardiac abnormalities (e.g. heart failure, arrhythmias, ischemic tachycardia, S-T segment deviations, etc.) from history or from cardiac stress testing in subjects ≥ 40 years old.
* Pneumonia
* Hepatic Failure/Jaundice
* Creatinine greater than 1.6 mg/dl
* Acute Cerebrovascular/ Neurological deficit
* Fever greater than 38 °C

Screening Laboratory Tests Exclusion Criteria

* Hematocrit lower than 32
* WBC lower than 3 thou/ul or greater than 14 thou/ul
* Liver Function Tests: SGOT and SGPT greater than twice upper limit of normal range (i.e. greater than 80 U/L).
* TBil greater than 2 mg/dl
* Alkaline Phosphatase greater than 150U/L
* Positive HIV, Hep B, Hep C
* Hepatic transaminase > 2x normal

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12-19 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in the level of catecholamines in plasma | An average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N Davis, MBBS, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No